CLINICAL TRIAL: NCT00000666
Title: A Randomized Prospective Study of Pyrimethamine Therapy for Prevention of Toxoplasmic Encephalitis in HIV-Infected Individuals With Serologic Evidence of Latent Toxoplasma Gondii Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Prevention
Other Study IDs: CPCRA 001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Toxoplasmosis, Cerebral; HIV Infections
Keywords: Toxoplasmosis; AIDS-Related Opportunistic Infections; Pyrimethamine; Drug Evaluation; Encephalitis; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Toxoplasmosis, Cerebral; HIV Infections; Toxoplasmosis; AIDS-Related Opportunistic Infections; Encephalitis; Acquired Immunodeficiency Syndrome | interventions — Pyrimethamine

INTERVENTIONS:
Drug: Pyrimethamine

SUMMARY:
To evaluate pyrimethamine as a prophylactic agent against toxoplasmic encephalitis in individuals who are coinfected with HIV and latent Toxoplasma gondii.

Toxoplasmic encephalitis is a major cause of illness and death in AIDS patients. Standard treatment for toxoplasmic encephalitis is to combine pyrimethamine and sulfadiazine. Continuous treatment is necessary to prevent recurrence of the disease, but constant use of pyrimethamine/sulfadiazine is associated with toxicity. Clindamycin has been shown to be effective in treatment of toxoplasmic encephalitis in animal studies. This study evaluates pyrimethamine as a preventive treatment against toxoplasmic encephalitis (per 3/26/91 amendment, clindamycin arm was discontinued).

DETAILED DESCRIPTION:
Toxoplasmic encephalitis is a major cause of illness and death in AIDS patients. Standard treatment for toxoplasmic encephalitis is to combine pyrimethamine and sulfadiazine. Continuous treatment is necessary to prevent recurrence of the disease, but constant use of pyrimethamine/sulfadiazine is associated with toxicity. Clindamycin has been shown to be effective in treatment of toxoplasmic encephalitis in animal studies. This study evaluates pyrimethamine as a preventive treatment against toxoplasmic encephalitis (per 3/26/91 amendment, clindamycin arm was discontinued).

Patients are randomized to receive pyrimethamine or placebo three times a week. All patients must be on aerosolized pentamidine, trimethoprim / sulfamethoxazole (T/S), or dapsone for Pneumocystis carinii pneumonia prophylaxis. Patients will be evaluated bi-weekly for the first month and every other month thereafter for at least 24 months.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Prophylactic treatment for Pneumocystis carinii pneumonia with aerosolized pentamidine, dapsone, or trimethoprim / sulfamethoxazole.

Allowed:

* Most medications not specifically excluded.

Prior Medication:

Allowed:

* Antivirals.
* Antiretrovirals.

Patients:

* Must be HIV positive or have an AIDS-defining illness OR be at known risk for HIV infection and have a CD4 cell count < 200/mm3 and no other known immunosuppressive disease.
* Must have positive titer for Toxoplasma gondii.
* Must be or become a patient of a CPCRA physician.
* May participate in other clinical trials as long as there is no potential activity against Toxoplasma gondii or cross-toxicity among study drugs.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* History of ocular, pulmonary, or central nervous system (CNS) toxicity.
* CNS lesions.
* Neurologic deficits except peripheral neuropathy.
* Mild, moderate, severe, or end-stage AIDS dementia complex. Grade 3 or higher nausea and/or vomiting.
* Sensitivity to pyrimethamine.

Concurrent Medication:

Excluded:

* On-going therapy with clindamycin, fansidar, methotrexate, trimetrexate, spiramycin, azithromycin, clarithromycin, 566C80, and/or sulfa agents other than anti-PCP agents.

Patients with the following are excluded:

* History of ocular, pulmonary, or central nervous system (CNS) toxicity.
* CNS lesions or history of CNS lesions.
* Neurologic deficits except peripheral neuropathy.
* Mild, moderate, severe, or end-stage AIDS dementia complex. Grade 3 or higher nausea and/or vomiting.
* Sensitivity to pyrimethamine.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Study Completion 1992-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobson M, Study Chair; Besch CL, Study Chair
Locations (16):
- United States (16):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Hill Health Corp, New Haven, Connecticut
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Jacobson MA, Besch CL, Child C, Hafner R, Muth K, Deyton L. Clinical programs for clinical research on AIDS: description of a randomized prospective study of clindamycin versus pyrimethamine for prevention of Toxoplasma gondii infection. Eur J Clin Microbiol Infect Dis. 1991 Mar;10(3):195-8. doi: 10.1007/BF01964462. PMID 1676364
- [Background] Jacobson MA, Besch CL, Child C, Hafner R, Matts JP, Muth K, Wentworth DN, Deyton L. Toxicity of clindamycin as prophylaxis for AIDS-associated toxoplasmic encephalitis. Community Programs for Clinical Research on AIDS. Lancet. 1992 Feb 8;339(8789):333-4. doi: 10.1016/0140-6736(92)91649-s. PMID 1346413
- [Background] Jacobson MA, Besch CL, Child C, Hafner R, Matts JP, Muth K, Wentworth DN, Neaton JD, Abrams D, Rimland D, et al. Primary prophylaxis with pyrimethamine for toxoplasmic encephalitis in patients with advanced human immunodeficiency virus disease: results of a randomized trial. Terry Beirn Community Programs for Clinical Research on AIDS. J Infect Dis. 1994 Feb;169(2):384-94. doi: 10.1093/infdis/169.2.384. PMID 8106772